CLINICAL TRIAL: NCT00571090
Title: Evaluation of Thyroid Fine Needle Aspiration Biopsies: Prediction of Thyroid Cancer From Ultrasonographic Characteristics of Thyroid Nodules
Brief Title: Prediction of Thyroid Cancer From Ultrasonographic Characteristics of Thyroid Nodules
Status: Completed | Type: Observational
Sponsor: Istanbul Science University (Other)
Collaborators: Group Florence Nightingale (Other)
Responsible Party: Principal Investigator, Ahmet Selcuk Can, Associate Professor of Medicine, Istanbul Science University
Other Study IDs: B.30.2.IBU.0.01.00.00/511; 511 (Other: Istanbul Science University)
Record Dates: First submitted 2007-12-10; First posted 2007-12-11 (Estimated); Last update posted 2014-03-31 (Estimated); Status verified 2014-03

CONDITIONS: Thyroid Nodule
Keywords: Thyroid nodule; Biopsy, Fine-Needle
MeSH Terms: conditions — Thyroid Nodule

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Thyroid nodule: Subjects who present with thyroid nodules will be enrolled into the study. Euthyroid and hypothyroid subjects with a solitary thyroid nodule or multinodular goiter will be enrolled. For subjects with a suppressed TSH, a thyroid scan will be performed. Subjects with a hypoactive nodule in the thyroid scan and a low TSH will be enrolled.
  Interventions: Procedure: Thyroid ultrasonography

INTERVENTIONS:
Procedure: Thyroid ultrasonography — Ultrasound-guided thyroid fine-needle aspiration biopsy

SUMMARY:
The aim of this study is to identify which ultrasonographic feature or a combination of features is the best predictor of thyroid cancer in thyroid nodules.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with thyroid nodules over 10 mm in the longest diameter
* Euthyroid or hypothyroid subjects with a solitary thyroid nodule or multinodular goiter
* Subjects with a hypoactive nodule in the thyroid scan and a low TSH

Exclusion Criteria:

* Subjects with four or more thyroid nodules that are over 10 mm
* Subjects with low TSH and hyperactive nodule on thyroid scan

Ages: 15 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Endocrinology Clinic
Sampling Method: Probability Sample
Enrollment: 735 (Actual)
Dates: Start 2003-06; Primary Completion 2012-07 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
Thyroid cancer | one year

CONTACTS AND LOCATIONS:
Overall Officials: Ahmet Selcuk Can, MD, Principal Investigator — Istanbul Science University and Group Florence Nightingale
Locations (1):
- Group Florence Nightingale, Istanbul, Turkey (Türkiye)

REFERENCES:
- [Background] Can AS. Cost-effectiveness comparison between palpation- and ultrasound-guided thyroid fine-needle aspiration biopsies. BMC Endocr Disord. 2009 May 16;9:14. doi: 10.1186/1472-6823-9-14. PMID 19445710
- See also: Free research article from the data of this protocol — http://www.biomedcentral.com/1472-6823/9/14